CLINICAL TRIAL: NCT03944824
Title: The Effect of Intradialytic Resistance Exercises Using Resistance Bands With Exercise Physiologist Consultation on the Physical Function of People Undergoing Hemodialysis: a Proof of Concept Study
Brief Title: The Effect of Intradialytic Exercise on the Physical Function of People Undergoing Hemodialysis
Acronym: IDEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Satellite Healthcare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SH066IDEX
Record Dates: First submitted 2019-02-12; First posted 2019-05-10 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: End Stage Renal Failure on Dialysis; Frail Elderly Syndrome
Keywords: Intra-Dialytic Exercise; End Stage Renal Disease; Hemodialysis; Therabands; Exercise Physiologist
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: The investigators will recruit 25 patients who will receive the exercise plans and once weekly visits from the exercise physiologists. 25 patients will be control. All 50 patients will receive pre and post physical function testing.
Masking Description: No masking, patients and physicians will be aware of their study arm assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Intervention) Arm (Experimental): The 25 patients in this arm will receive an interventional exercise plan using resistance bands and once weekly visits from an exercise physiologist while on dialysis for 12 weeks. They will undergo a frailty screening using a Modified Fried Frailty Scale at the beginning and end of the trial to include: Timed up and Go test, Sit-to-Stand Test, Handgrip Strength Test, Low physical activity questionnaire.
  Interventions: Other: Exercise Plan using resistance bands; Diagnostic Test: Modified Fried Frailty Scale
- Control (Placebo Comparator): The 25 patients in the control arm will not receive an interventional exercise plan or visits from an exercise physiologist while on dialysis for 12 weeks. They will undergo a frailty screening using a Modified Fried Frailty Scale at the beginning and end of the trial to include: Timed up and Go test, Sit-to-Stand Test, Handgrip Strength Test, Low physical activity questionnaire.
  Interventions: Diagnostic Test: Modified Fried Frailty Scale

INTERVENTIONS:
Other: Exercise Plan using resistance bands — Exercise under the guidance of an exercise physiologist using elastic resistance bands and weekly meeting with an exercise physiologist for 12 weeks
  Arms: Exercise (Intervention) Arm
Diagnostic Test: Modified Fried Frailty Scale — Patients will be screened for frailty pre and post with sit-to-stand test, timed up and go test, handgrip strength test and administered the low physical activity questionnaire. These components together consist of the Modified Fried Frailty Index.

SUMMARY:
The investigators intend to recruit 50 patients into an intradialytic exercise study that will measure the impact of resistance bands exercises under the guidance of an exercise physiologist on the physical function of hemodialysis patients.

DETAILED DESCRIPTION:
The primary objective of this study will be to test the feasibility and efficacy of a 3 month exercise physiologist consultation program. Specifically, the investigator's aims will be to:

1. Test the feasibility of a 3-month exercise physiologist led program
2. Measure the effect of an exercise physiologist collaboration and intradialytic exercise on the physical function of HD patients using the 30 second STS test, handgrip strength test [required for frailty scale], 8-foot TUG test and patient physical activity based off of the Low Physical Activity Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Ability to understand and communicate English
* Diagnosis of ESRD and currently undergoing in-center hemodialysis
* On HD for longer than 6 weeks
* Approved by the Satellite Milpitas Medical Director and/or referring physician

Exclusion Criteria:

* Previous major amputations
* Inability to independently ambulate
* Known to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Rate of Patient Adherence to Exercise Regimen | 12 weeks
  Adherence calculated as the total number of self-reported exercise sessions attempted by the patient when EP not present divided by the total number of hemodialysis sessions.
Rate of Adverse Events Secondary to Exercises | 12 weeks
  Adverse events defined as any injury, impairment or medical condition that was directly or suspected to be due to performing the prescribed exercise. This information will be collected from the patient at the weekly meeting with the EPs.

SECONDARY OUTCOMES:
Change in Sit-To-Stand Test | 12 weeks
  Change in physical function as measured by the 30 second sit to stand test (STS)
Change in Handgrip Strength Test | 12 weeks
  Change in handgrip strength following the 12 week intervention as measured by a handgrip dynanometer
Change in Timed Up and Go Test | 12 weeks
  Change in 8 foot timed up and go test (TUG).

CONTACTS AND LOCATIONS:
Locations (1):
- Satellite Milpitas, Milpitas, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Bao Y, Dalrymple L, Chertow GM, Kaysen GA, Johansen KL. Frailty, dialysis initiation, and mortality in end-stage renal disease. Arch Intern Med. 2012 Jul 23;172(14):1071-7. doi: 10.1001/archinternmed.2012.3020. PMID 22733312
- [Background] McAdams-DeMarco MA, Law A, Salter ML, Boyarsky B, Gimenez L, Jaar BG, Walston JD, Segev DL. Frailty as a novel predictor of mortality and hospitalization in individuals of all ages undergoing hemodialysis. J Am Geriatr Soc. 2013 Jun;61(6):896-901. doi: 10.1111/jgs.12266. Epub 2013 May 27. PMID 23711111
- [Background] Johansen KL, Delgado C, Kaysen GA, Chertow GM, Chiang J, Dalrymple LS, Segal MR, Grimes BA. Frailty Among Patients Receiving Hemodialysis: Evolution of Components and Associations With Mortality. J Gerontol A Biol Sci Med Sci. 2019 Feb 15;74(3):380-386. doi: 10.1093/gerona/gly206. PMID 30192916
- [Background] Heiwe S, Jacobson SH. Exercise training for adults with chronic kidney disease. Cochrane Database Syst Rev. 2011 Oct 5;2011(10):CD003236. doi: 10.1002/14651858.CD003236.pub2. PMID 21975737
- [Background] Cho JH, Lee JY, Lee S, Park H, Choi SW, Kim JC. Effect of intradialytic exercise on daily physical activity and sleep quality in maintenance hemodialysis patients. Int Urol Nephrol. 2018 Apr;50(4):745-754. doi: 10.1007/s11255-018-1796-y. Epub 2018 Jan 23. PMID 29362960
- [Background] Guio BM, Gomes CP, Costa FBD, Oliveira ADS, Duarte MT, Leite M Junior. Beneficial effects of intradialytic cardiopulmonary rehabilitation. J Bras Nefrol. 2017 Jul-Sep;39(3):275-282. doi: 10.5935/0101-2800.20170051. English, Portuguese. PMID 29044337
- [Background] Young HML, March DS, Graham-Brown MPM, Jones AW, Curtis F, Grantham CS, Churchward DR, Highton P, Smith AC, Singh SJ, Bridle C, Burton JO. Effects of intradialytic cycling exercise on exercise capacity, quality of life, physical function and cardiovascular measures in adult haemodialysis patients: a systematic review and meta-analysis. Nephrol Dial Transplant. 2018 Aug 1;33(8):1436-1445. doi: 10.1093/ndt/gfy045. PMID 29608708
- [Background] Gomes Neto M, de Lacerda FFR, Lopes AA, Martinez BP, Saquetto MB. Intradialytic exercise training modalities on physical functioning and health-related quality of life in patients undergoing maintenance hemodialysis: systematic review and meta-analysis. Clin Rehabil. 2018 Sep;32(9):1189-1202. doi: 10.1177/0269215518760380. Epub 2018 Feb 26. PMID 29480025
- [Background] Bennett PN, Fraser S, Barnard R, Haines T, Ockerby C, Street M, Wang WC, Daly R. Effects of an intradialytic resistance training programme on physical function: a prospective stepped-wedge randomized controlled trial. Nephrol Dial Transplant. 2016 Aug;31(8):1302-9. doi: 10.1093/ndt/gfv416. Epub 2015 Dec 28. PMID 26715763
- [Background] Anding K, Bar T, Trojniak-Hennig J, Kuchinke S, Krause R, Rost JM, Halle M. A structured exercise programme during haemodialysis for patients with chronic kidney disease: clinical benefit and long-term adherence. BMJ Open. 2015 Aug 27;5(8):e008709. doi: 10.1136/bmjopen-2015-008709. PMID 26316654
- [Background] Bennett PN, Peter J, Wang W, Street M. Attitudes of Nephrology Nurses Toward Patient Exercise During Hemodialysis. Nephrol Nurs J. 2016 Jul-Aug;43(4):331-337. PMID 30550060
- [Background] Bennett PN, Daly RM, Fraser SF, Haines T, Barnard R, Ockerby C, Kent B. The impact of an exercise physiologist coordinated resistance exercise program on the physical function of people receiving hemodialysis: a stepped wedge randomised control study. BMC Nephrol. 2013 Sep 27;14:204. doi: 10.1186/1471-2369-14-204. PMID 24070232
- [Background] Johansen KL, Painter P, Delgado C, Doyle J. Characterization of physical activity and sitting time among patients on hemodialysis using a new physical activity instrument. J Ren Nutr. 2015 Jan;25(1):25-30. doi: 10.1053/j.jrn.2014.06.012. Epub 2014 Sep 8. PMID 25213326

DOCUMENTS (2):
  • Informed Consent Form (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/24/NCT03944824/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT03944824/Prot_SAP_001.pdf